CLINICAL TRIAL: NCT06316700
Title: A Pharmacokinetic Study of a Novel Nutritional Product on Healthy Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: AG-02-0124
Record Dates: First submitted 2024-02-21; First posted 2024-03-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Powder Supplement (Active Comparator): A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Interventions: Dietary Supplement: Nutritional supplement
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Arms: Nutritional Powder Supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=16 apparently healthy men and women. The purpose of this study is to examine the bioavailability of a health and wellness supplement.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 18 and 45 yr (inclusive).
* Body Mass Index of 18.5-29.9 (inclusive).
* Body weight of at least 120 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate and record their previous 24-hour diet, refrain from caffeine and exercise for 24 hours prior to each visit, and fast for 10 hours prior to each visit.
* Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
* Subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* Multivitamin/Multimineral supplement consumption within the past 3 months
* Additionally, eligible participants cannot regularly consume (i.e., at least five days/week) resveratrol, quercetin, pterostilbene, coQ10, grapefruit, nicotinamide riboside, probiotics, prebiotic fiber, green tea, niacin (vitamin B3), multivitamin/multimineral, or products meant to promote "healthy aging" or "anti-aging" or "longevity" products in the 2 months prior to screening as well as throughout the study.
* Subjects who have received an antibiotic, antifungal, antiparasitic, or antiviral treatment within 3 months prior to study entry.
* History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* History of use of medications (e.g., Retinoids, levodopa, statins, loop diuretics) or dietary supplements known to confound the study or its endpoints.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
* Current smokers, vapers, or tobacco users or use of tobacco within the past month.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc.
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, Inflammatory bowel syndrome (IBS), Inflammatory bowel disease (IBD; e.g., Crohn's, ulcerative colitis), diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition (e.g., rheumatoid arthritis, , Lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women. Women who participate in this study must agree to the use of contraception for the duration of the study and any woman that is sexually active will have to take pregnancy test prior to enrolling with a negative result. Women of childbearing age (any woman prior to menopause) regardless of their use of contraception will be provided a urine pregnancy test kit at their screening visit and take the test in private using the female lavatory after signing an informed consent.
* A change in hormone therapy, including oral contraceptives, within 4 weeks prior to screening, or unwilling to maintain current hormone therapy/oral contraceptive use throughout the course of the study.
* Known sensitivity to any ingredient in the test formulations as listed in the product label.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.
* Subject is engaged in a specialty diet including but not limited to, Vegan, Vegetarian, Ketogenic, Paleo, Atkins, South Beach, Carnivore, etc.
* Subjects that have donated blood or plasma within the previous week.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of zinc following consumption of study products | Baseline & 30, 60, 90, 120, 180, 240, 360, 480 minutes post-ingestion
  Zinc (ug/dl)
Plasma concentration of Vitamin C following consumption of study products | Baseline & 30, 60, 90, 120, 180, 240, 360, 480 minutes post-ingestion
  Vitamin C (mg/dl)
Plasma concentration of Folate following consumption of study products | Baseline & 30, 60, 90, 120, 180, 240, 360, 480 minutes post-ingestion
  Folate (ng/ml)
Plasma concentration of calcium following consumption of study products | Baseline & 30, 60, 90, 120, 180, 240, 360, 480 minutes post-ingestion
  Calcium (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No